CLINICAL TRIAL: NCT05831501
Title: Postoperative Analgesic Efficacy of Trans Abdominis Plane Block in Women Undergoing Caesarean Section, a Randomized Controlled Trial
Brief Title: Postoperative Analgesic Efficacy of Trans Abdominis Plane Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, clinical professor, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IERB/02/2023
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Post Operative Pain; Cesarean Section Complications
Keywords: TAP block, C-section, Spinal anesthesia, localized field effects, analgesia, Postoperative pain and Opioids
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block group (Experimental): At the end of the cesarean section, a TAP block will be given by Injecting of 20ml 0.25% Bupivacaine on both sides of the midline using ultrasound-guided subcostal approach
  Interventions: Procedure: Trans abdominis plane block
- Placebo group (No Intervention): At the end of the cesarean section, 20 ml of saline will be injected on both sides of the midline

INTERVENTIONS:
Procedure: Trans abdominis plane block — Ultrasound guided infiltration of local anaesthetic bupivacaine via 22G Quincke needle between internal oblique and trans abdominis muscle layers in abdominal wall.
  Arms: TAP block group

SUMMARY:
Transverse abdominis plane (TAP) block is an effective method to manage postoperative pain in patients with midline abdominal wall incisions. It is used frequently in many lower abdominal surgeries however its use after caesarean section is still new, and fewer studies are available. We conducted this study to see the analgesic effect of TAP block after caesarean section.

DETAILED DESCRIPTION:
The study is being conducted, at Combined Military Hospital Sargodha, Pakistan, to compare the analgesic efficacy of TAP block in providing post-caesarean analgesia with the control group, in terms of mean postoperative use of opioids after caesarean delivery. Sixty patients have been randomly selected using non-probability, consecutive sampling, and applying inclusion and exclusion criteria. The study design is a randomized controlled trial with thirty patients in each group undergoing elective caesareans. All patients will be given spinal anaesthesia with 1.5ml of 0.75% hyperbaric bupivacaine for a caesarean section. Patients in Group A will receive bilateral TAP block with 20ml of 0.25% bupivacaine while 20 ml of saline will be injected in patients of Group B on both sides of midline after caesarean section, in addition to intravenous ketorolac 8hrly. The intensity of pain, total opioid consumption, presence of vomiting, and sedation will be noted until 24 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective Caesarean section
* ASA 1-3
* 20yrs to 45yrs

Exclusion Criteria:

* Emergency Surgery
* known allergy to local anaesthetic
* severe pre-eclampsia
* placenta accreta
* ASA 4
* Coagulopathy
* Hemodynamically unstable

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 24 hours post cesarean section
  within 24hours after surgery

SECONDARY OUTCOMES:
Pain intensity Score | from end of secarean section till 24 post operative hours
  Pain intensity at 6 hours,12 hours and 24 hours after surgery
Vomiting | Within 24hours after surgery
  frequency of vomiting within 24hours after surgery
Duration of First Rescue Analgesia | Within 24hours after surgery
  time after surgery when first dose of opioid required

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Military Hospital, Sargodha, Punjab Province, Pakistan